CLINICAL TRIAL: NCT01319279
Title: An Open-Label, Single-Dose, Parallel-Group Study to Assess the Pharmacokinetics of the Hydrocodone Bitartrate Extended-Release Tablet (15 mg) in Subjects With Normal Hepatic Function and Subjects With Moderate Hepatic Impairment
Brief Title: A Study to Evaluate the Pharmacokinetics of the Hydrocodone Extended-Release Tablet (CEP-33237) in Subjects With Normal Hepatic Function and Subjects With Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C33237/1089
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Hepatic Impairment
Keywords: Pharmacokinetics; Hydrocodone; Extended Release; Hepatic impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Hepatic Function (Experimental): Intervention Drug: Hydrocodone bitartrate extended-release tablet
  Interventions: Drug: Hydrocodone bitartrate extended-release tablet
- Moderate Hepatic Impairment (Experimental): Intervention Drug: Hydrocodone bitartrate extended-release tablet
  Interventions: Drug: Hydrocodone bitartrate extended-release tablet

INTERVENTIONS:
Drug: Hydrocodone bitartrate extended-release tablet — 15 mg (single dose)

SUMMARY:
The purpose of this study is:

1. To assess the pharmacokinetics of the hydrocodone bitartrate extended-release tablet in subjects with moderate hepatic impairment and in subjects with normal hepatic function.
2. To assess the safety and tolerability of the hydrocodone bitartrate extended-release tablet in subjects with moderate hepatic impairment and in subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects:

   * Written informed consent is obtained
2. Subjects with normal hepatic function:

   * The subject is in generally good health (age-appropriate) as determined by medical and psychiatric history, physical examination, ECG, serum chemistry, hematology, coagulation, urinalysis, and serology.
3. Subjects with hepatic impairment:

   * The subject's health is otherwise clinically stable as determined by medical history, physical examination, ECG, serum chemistry, hematology, coagulation parameters (PT, activated partial thromboplastin time [aPTT], and international normalized ratio [INR]), urinalysis, and serology except for those signs and symptoms attributable to liver disease.
   * The subject has case record notes demonstrating physical signs consistent with 1 or more of the following characteristic clinical manifestations of liver cirrhosis: liver firmness to palpation, splenic enlargement, spider angiomas, palmar erythema, parotid hypertrophy, testicular atrophy, ascites (accumulation of fluid in the abdominal cavity), or gynecomastia.
   * The subject has a Child-Pugh Classification score of 7-9 points (moderate).

Exclusion Criteria:

1. All subjects:

   * The subject has any clinically significant, uncontrolled medical condition.
   * The subject is a poor metabolizer of CYP2D6 substrates based on genotyping performed at screening.
   * The subject has previously participated in a study with CEP-33237.
   * The subject has a known sensitivity or idiosyncratic reaction to hydrocodone or hydromorphone, related compounds, or to any metabolites, or any compound listed as being present in a study formulation.
2. Subjects with normal hepatic function:

   * The subject has a positive test result for HBsAg or antibodies to hepatitis C.
   * The subject has a history of alcohol, narcotic, or any other substance abuse.
3. Subjects with hepatic impairment:

   * The subject has severe ascites.
   * The subject has an acute exacerbation of liver disease as indicated by worsening clinical signs of hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC and Cmax) after a single dose | 7 days

SECONDARY OUTCOMES:
Safety (occurrence of adverse events, labs, ECG, physical exam, vital signs, oxygen saturation) | throughout the 37 day study period (includes screening, drug administration and pharmacokinetics sampling period, and follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon, Inc.
Locations (1):
- Orlando Clinical Research, Orlando, Florida, United States